CLINICAL TRIAL: NCT06758505
Title: Rehabilitation Strategies for Social Participation in Chronic Stroke Survivors
Acronym: START2ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Minmei Shih, Research Scientist, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY24030133; R03HD114635 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2025-01-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Chronic Phase of Disease
Keywords: Strategy Training; Acceptance and Commitment Therapy; Social Participation
MeSH Terms: conditions — Stroke | interventions — N-(2-acetamido)-2-aminoethanesulfonic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACES (Experimental)
  Interventions: Behavioral: Strategy Training embedded with Acceptance and Commitment Therapy Principles
- START (Active Comparator)
  Interventions: Behavioral: Strategy Training Only

INTERVENTIONS:
Behavioral: Strategy Training Only — Participants will receive ten 45-60-minute sessions (two times per week) in person in their residence to address real-world performance with an emphasis on START strategy, task-specific practice, and guided discovery to perform social participation activities. In session 1, participants will be guided to select 3 to 5 meaningful social activities and prioritize them. In sessions 2 - 9, participants will use structured START strategy worksheet to try the selected activity; assess execution (e.g., what went well, what did not); reflect on a plan with specific strategies and to address identified challenges; and try social participation activities again. The interventionist will use guided discovery to support START strategy application and to elicit problem solving skills. This process will be repeated iteratively across sessions. In session 10, participants will summarize lessons learned and generate an action plan for after the intervention.
  Other Names: START
  Arms: START
Behavioral: Strategy Training embedded with Acceptance and Commitment Therapy Principles — Participants will receive ten 45-60-minute sessions (two times per week) in person in their residence to address real-world performance with task-specific practice and an emphasis on psychological processes using ACT principles. In session 1, participants will clarify value-consistent social participation goals for engaging in 3-5 meaningful activities ("Do What Matters"). In sessions 2-9, participants will be guided applying ACT principles to cope with negative experiences and separate self from thoughts and feelings ("Open Up") and practice mindfulness, stimulate awareness, recognize same person with different experiences, and build self-compassion ("Be Present"). This process (i.e., try an activity that aligns with values and committed actions; assess performance; and reflect on a plan) will be repeated iteratively. In session 10, participants reflect on lessons learned and generate an action plan for after the intervention.
  Other Names: ACES
  Arms: ACES

SUMMARY:
The goal of this clinical trial is to test a new rehabilitation program, combining acceptance and commitment therapy with strategy training (ACES), to help people resume social participation after stroke and live in the community.

Investigators will also compare the changes in social participation and psychological flexibility from baseline to follow-up at one-month after rehabilitation to see if participants who receive ACES report clinically meaningful improvements (Cohen's d=0.2 or greater) compared to the existing rehabilitation program using strategy training alone (START).

Participants will:

* complete testing to see if they are eligible for the study. If qualified, complete testing to understand how the stroke has affected their daily life
* be randomized to receive either ACES or START rehabilitation program for 10 sessions at their home
* repeat part of the tests at the end of the intervention and one month after

DETAILED DESCRIPTION:
In April 2025, the investigator changed the recruitment status because the first enrolled participant ended up being ineligible. The investigators also updated eligibility criteria and outcome measures to be consistent with the IRB protocol.

In June 2025, the investigator received notice of award from NIH and thus updated information to be consistent with the IRB protocol.

ELIGIBILITY:
Inclusion Criteria:

1. primary diagnosis of chronic stroke, ≥6 months post onset,
2. ≥18 years old,
3. community-dwelling (i.e., living in a residential setting in the community),
4. restrictions in social participation, indicated by Activity Card Sort (<80% of pre-stroke activities)

Exclusion Criteria:

1. progressive neurological diagnosis (e.g., dementia, Parkinson's disease, multiple sclerosis, or brain tumor) reported by participants or proxy,
2. inability to provide written informed consent,
3. severe aphasia (score 0 or 1 on the Boston Diagnostic Aphasia Examination 3rd Edition Severity Rating Scale),
4. currently undergoing stroke rehabilitation or mental health intervention (but participation in maintenance sessions, self-help groups, or couples therapy is permitted),
5. major depressive disorder, indicated by PRIME-MD, unless undergoing treatment for at least 4 weeks and are released to participate by their physician or counselor
6. bipolar or psychotic disorder, indicated by PRIME-MD, or
7. substance use disorder within 3 months, indicated by Mini-International Neuropsychiatric Interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Fidelity (for each group) | Baseline to Post-intervention up to 8 weeks
  Fidelity is measured using Strategy Training (ST) and Acceptance and Commitment Therapy (ACT) fidelity tools.
  All intervention sessions will be video recorded and a random 20 percent will be rated by independent evaluators trained by the principal investigator. ST fidelity will be assessed with the 10-item fidelity tool with 8 or more items rated as adequate or excellent indicating adequate fidelity. ACES fidelity will be assessed with a 22-item tool generated from the 10-item ST and 12-item ACT fidelity tools, with 18 or more items rated as adequate or excellent indicating adequate fidelity. The a priori criterion for adequate fidelity was that equal or greater than 80 percent of intervention sessions are rated with equal or greater than 80 percent of adequate fidelity for each START and ACES intervention.
Feasibility: Satisfaction (for each group) | Baseline to Post-intervention up to 8 weeks
  Client satisfaction is measured using the Client Satisfaction Questionnaire. The Clients Satisfaction Questionnaire is an 8-item assessment of satisfaction with the intervention program, rated on a 4-point scale that ranges from 1 to 4 in each item. An average score will be computed for each participant. High scores indicate high satisfaction. The a priori criterion for satisfaction was equal or greater than 80 percent of the sample has mean Client Satisfaction Questionnaire score of equal or greater than 2.5.

SECONDARY OUTCOMES:
Changes in social participation: Difficulty to participate in social activities | Baseline to 1- Month Post-intervention (Follow-up) up to 12 weeks
  Changes in social participation measured by PROMIS Ability to Participation in Social Roles and Activities.
  The PROMIS Ability to Participate in Social Roles and Activities (APS) is a self-report measure that assesses difficulty participation in social roles and activities. APS is an 8-item short form rated on a 5-point scale. High scores indicate high difficulty. The total raw score will be transformed into a t-score that ranges from 0 to 100, with a mean of 50 and a standard deviation of 10.
  The a priori criterion for change was a small effect size of change (d=0.2 or greater).
Changes in social participation: Satisfaction with social participation | Baseline to 1- Month Post-intervention (Follow-up) up to 12 weeks
  Changes in social participation measured by PROMIS Satisfaction with Social Roles and Activities.
  The PROMIS Satisfaction with Social Roles and Activities (SPS) is a self-report measure that assesses satisfaction with participation in social roles and activities. SPS is 8-item short form rated on a 5-point scale. High scores indicate low satisfaction. The total raw score will be transformed into a t-score that ranges from 0 to 100, with a mean of 50 and a standard deviation of 10.
  The a priori criterion for change was a small effect size of change (d=0.2 or greater).
Changes in psychological flexibility | Baseline to 1- Month Post-intervention (Follow-up) up to 12 weeks
  Changes in psychological flexibility measured by Multidimensional Psycho-logical Flexibility Inventory.
  The Multidimensional Psycho-logical Flexibility Inventory (MPFI) is a self-report measure that assesses psychological flexibility and psychological inflexibility. Each psychological flexibility and inflexibility domain includes 6 scales and each scale has 5 items, rated on a 6-point scale. A total score will be computed for each psychological flexibility and inflexibility domain that ranges from 6 to 180. High scores indicate high levels of measured psychological flexibility and psychological inflexibility.
  The a priori criterion for change was a small effect size of change (d=0.2 or greater).
Changes in wellbeing | Baseline to 1- Month Post-intervention (Follow-up) up to 12 weeks
  Changes in wellbeing measured by Veterans RAND 12-item Health Survey. The Veterans RAND 12-item Health Survey (RAND-12) is a self-report measure that assesses wellbeing ranging from physical to mental health. Items rated on a 5-point scale. Results are summarized as physical component score (PCS) and mental component score (MCS). The raw scores of the PCS and MCS will be transformed into Z-scores that range from 0 to 100, with a mean of 50 and a standard deviation of 10. High scores indicate high levels of wellbeing.
  The a priori criterion for change was a small effect size of change (d=0.2 or greater).

CONTACTS AND LOCATIONS:
Overall Officials: Minmei Shih, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No